CLINICAL TRIAL: NCT00366353
Title: A Randomized Trial Comparing Sedation Versus No Sedation For Patients Undergoing a Spontaneous Breathing Trial.
Brief Title: Sedation Versus No Sedation in a Spontaneous Breathing Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty obtaining enrollment
Sponsor: Memorial Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 05-10
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Respiratory Insufficiency
Keywords: Mechanical Ventilation; Spontaneous Breathing Trial; Sedation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Sedation suring a spontaneous breathing trial.
  Interventions: Other: Sedation during SBT
- 2 (Other): No sedation during spontaneous breathing trial
  Interventions: Other: No sedation

INTERVENTIONS:
Other: Sedation during SBT
  Arms: 1
Other: No sedation
  Arms: 2

SUMMARY:
An important part of how we decide when a patient is ready to have their breathing tube removed is to have a person breathe without any machine breaths while the breathing tube is still in place. We call this a spontaneous breathing trial.

Commonly, while patients have the breathing tube, they are given medications to keep them sedated and comfortable so breathing does not bother them. These medicines are often stopped before the spontaneous breathing trial so they can be more awake for the test.

There are signs the doctors look for during the spontaneous breathing trial that suggest the patient might not be ready for the breathing trial to come out. Signs like fast breathing, small breaths, a fast heart rate, or looking more anxious than usual may mean that the patient is not ready to come off the ventilator. However, if someone has been given sedation medicines the entire time they have had a breathing tube and are then woken up, they may naturally get very anxious. They may show the same signs as someone who is failing their breathing test, but in their case these signs are only because they are anxious.Doctors may mistake these signs as failing the breathing test and may not pull the breathing tube out even though the patient is really ready for it to come out.

We wish to try and find out if patients do better during their spontaneous breathing trials if they are continued on some sedative medicines to treat anxiety or if they do better if the medicines are stopped before the test.

DETAILED DESCRIPTION:
All intubated patients cared for by the Medical Intensive Care Unit (MICU)team during the study period will be evaluated. After 24 hours of mechanical ventilation, patients not meeting any exclusionary criteria will be considered for entrance into our trial. We will attempt to obtain consent as soon as the 24 hour period is fulfilled, even if the patient is not ready for extubation at that point. This is to maximize the success rate for obtaining consent without delaying the SBT when the patient is clinically ready. Given the nature of this protocol, we expect that the informed consent will primarily be obtained from the patient's family member or POA. For all patients who regain competency, they will be re-consented for permission to use their data that has been collected.

Once patients are consented, they will be followed daily by the study investigators. When the order is written by the MICU team for the patient to undergo a SBT, the patient's level of consciousness will be evaluated by the nursing staff using the RASS. If the patient's score is <(-2), they will notify the study investigators. The patient will then be randomized by sealed envelope to one of two study groups. Group 1 will immediately undergo their SBT while still sedated. Group 2 will have their sedation held. Once their RASS score is 0 or higher and they can follow simple commands (holding up two fingers to command), they will be initiated on their SBT.

The standard duration of an SBT by protocol is 2 hours. The duration of SBT may be shorter at the discretion of the ICU attending physician. Additionally, the standard ventilators settings for an SBT is 10 cm of Pressure Support and 5 cm of PEEP (positive and expiratory pressure). This may vary some by the attending's preference though we encourage the use of the standard setting during the study unless there is a clear need to deviate from the protocol. This is to limit the confounding impact that differing levels of Pressure Support may have on the parameters tracked. Patients who are felt to be failing the SBt will be placed back on fill ventilator support at any point directed by the MICU team. Given the lack of objective criteria to define failure of SBT, there are no clear criteria defined and the decision that a patient is failing their SBT will be determined by the attending physician.

Nursing staff will be provided with a documentation form (Data sheet 1) and asked to annotate heart rate, blood pressure, respiratory rate, tidal volume, oxygen saturation, and RASS score at 0, 15, 30, 60 minutes and at the conclusion of the SBT.They will be inserviced on the protocol prior to the start of the study. The study investigators will collect demographic information and record it on Data sheet 2. In addition to the primary endpoint(changes in cardiopulmonary parameters and RASS collected by the nursing staff), secondary endpoints will include outcome of first SBT(pass or fail), time from randomization to extubation, outcome of the first extubation (Data sheet 1). As stated earlier, there are no clearly defined cut-off values for any of the monitored variables that define failure of an SBT.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 or older
* Intubation time greater than or equal to 24 hours
* Patient is sedated at the time the MICU writes the order for the SBT. A RASS score of less than -2 will be considered sedated

Exclusion Criteria:

* Acute brain injury
* Pregnancy
* Wards of the state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Changes in cardiopulmonary variables and RASS during the SBT | 2hrs unless directed by ICU attending physician

SECONDARY OUTCOMES:
Time from randomization to the first SBT | Time of first SBT

CONTACTS AND LOCATIONS:
Overall Officials: Jack L DePriest, Principal Investigator — Memorial Medical Center
Locations (1):
- Memorial Medical Center, Johnstown, Pennsylvania, United States